CLINICAL TRIAL: NCT04984109
Title: The Effect of Preoperative Ultrasound-guided Pericapsular Nerve Group Block (PENG) on the Postoperative Analgesia After Total Hip Arthroplasty: Randomized Controlled Study
Brief Title: Ultrasound-guided PENG Block in Total Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sameh Abdelkhalik Ahmed Ismaiel, Assistant Professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 34582/3/21
Record Dates: First submitted 2021-07-24; First posted 2021-07-30 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Pain, Postoperative; Opioid Overdose
Keywords: Hip arthroplasty; Pericapsular nerve block; Pain
MeSH Terms: conditions — Pain, Postoperative; Opiate Overdose; Pain

STUDY DESIGN:
Intervention Model Description: Prospective study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: * Sham ESP block will be administrated in the control group
  * Measurements will be obtained by anesthetists not participating in the study and blinded to its group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): Patients will receive preoperative US-guided will receive sham PENG with an injection of just 1mL saline.
  Interventions: Procedure: Sham PENG block
- PENG Group (Experimental): Patients will receive preoperative US-guided will receive real PENG with an injection of 20mL of bupivacaine 0.25%+ 0.2mg/mL dexamethasone.
  Interventions: Procedure: Real PENG block

INTERVENTIONS:
Procedure: Sham PENG block — The regional block will be performed with the patient in the supine position in operative area with adequate groin exposure. The probe will first be placed at the anterior superior iliac spine in transverse plane, and then will be moved caudally to identify anterior inferior iliac spine (AIIS). The probe will be then rotated to align the AIIS and iliopubic eminence (IPE). This will reveal the iliopsoas tendon and muscle together with femoral vessels superficially. A 22-G 100-mm echogenic needle will be inserted in-plane from lateral to medial, and the tip will be kept at the midpoint of AIIS and IPE deep to psoas tendon. After lifting of psoas tendon by hydrolocation, the patients in PENG group will receive 1 mL of normal saline.
  Arms: Control group
Procedure: Real PENG block — The regional block will be performed with the patient in the supine position in operative area with adequate groin exposure. The probe will first be placed at the anterior superior iliac spine in transverse plane, and then will be moved caudally to identify anterior inferior iliac spine (AIIS). The probe will be then rotated to align the AIIS and iliopubic eminence (IPE). This will reveal the iliopsoas tendon and muscle together with femoral vessels superficially. A 22-G 100-mm echogenic needle will be inserted in-plane from lateral to medial, and the tip will be kept at the midpoint of AIIS and IPE deep to psoas tendon. After lifting of psoas tendon by hydrolocation, the patients in PENG group will receive 20 ml of (0.25%) bupivacaine with 0.2 mg/mL dexamethasone that will be injected in 5 ml aliquots after negative aspiration.
  Arms: PENG Group

SUMMARY:
* This randomized controlled study will be carried out on 60 adult patients undergoing primary total hip replacement in Tanta University Hospitals. All Patients will receive spinal anesthesia with either sham or real US-guided PENG block.
* The primary outcome will be the time to first request for rescue analgesia. The secondary outcome will be the postoperative Numeric Rating Scale (NRS) score and the total morphine consumption (rescue analgesia) in the first 24 h postoperatively.

DETAILED DESCRIPTION:
* This prospective randomized double-blinded study will be carried out on 60 adult patients admitted to Tanta University Hospitals for 6 months started immediately after approval of the Institutional Ethical Committee.
* A written informed consent will be obtained from each patient. All data of patients will be confidential with secret codes and private files for each patient, all given data will be used for scientific purposes only after an explanation of the purpose of the study to all patients. - Any unexpected risks encountered during the course of the research will be cleared to the patients as well as to the ethical committee on time.
* The primary endpoint is a prolongation of the postoperative analgesia and reduction of the postoperative analgesic consumption. The study will be terminated if local anesthetic toxicity occurs and this will be announced to the participants and to the ethical committee at the time and adequate measures will be taken to resolve and avoid these risks.
* Group allocation will be done by using computer-generated software of randomization introduced into sealed opaque envelope technique. A blinded nurse, who does not participate in the study or data collection, will read the number contained in the envelope and make group assignments. All the nerve blocks will be performed by one anesthesiologist.

  * Control Group: (30 patients) will receive sham PENG (just 1mL saline)
  * PENG Group: (30 patients) will receive real PENG (20mL of bupivacaine 0.25% plus 0.2mg/ml dexamethasone)

Anesthetic technique:

•Preoperative assessment will be done by: History taking. Clinical examination. Laboratory investigations including complete blood count, bleeding and clotting times, APTT, liver and kidney function tests.

During the pre-anesthetic assessment, all patients will be familiarized with the Numeric Rating Scale (NRS) score.

* In the holding area, After the establishment of intravascular access by introducing an 18-gauge intravenous (IV) cannula, all the patients will be preloaded with Ringer's lactate solution (7 mL/kg).
* On arrival at operation room, Routine monitoring of heart rate by ECG, noninvasive blood pressure (NIBP), pulse oximetry will be done.

  * Lumbar puncture will be performed at the level of L3-L4/L4-L5 intervertebral space with a 25-gauge spinal needle. After ensuring free flow of cerebrospinal fluid, 2 mL of hyperbaric bupivacaine solution (0.5%) (10mg)) with 0.5 mL (25 µg) fentanyl will be injected. The sensory block will be assessed by loss of sensation to pinprick test. The level of the sensory block should achieve at least a level of T10. Moreover, the motor block will be assessed by modified Bromage score till reaching at least a score of 2. (0; means the ability of the patient to move the hip, knee, and ankle, 1; means the inability of the patient to move the hip, but can move the knee and ankle, 2; means the inability of the patient to move the hip and knee, but can move the ankle, and finally 3; means the inability of the patient to move the hip, knee, and ankle). If the sensory and motor block levels will not be achieved within 20 minutes, the patient will be excluded from the study and receive general anesthesia. If the sensory and motor block will be achieved, the patient will receive an ultrasound-guided PENG block before starting the surgery.
  * ThePENG block will be performed with the patient in the supine position in the operative area with adequate groin exposure. The probe will first be placed at the anterior superior iliac spine in the transverse plane, and then will be moved caudally to identify the anterior inferior iliac spine (AIIS). The probe will be then rotated to align the AIIS and iliopubic eminence (IPE). This will reveal the iliopsoas tendon and muscle together with femoral vessels superficially. A 22-G 100-mm echogenic needle will be inserted in-plane from lateral to medial, and the tip will be kept at the midpoint of AIIS and IPE deep to psoas tendon. After lifting of the psoas tendon by hydrolocation, the patients in the PENG group will receive 20 ml of (0.25%) bupivacaine with 0.2 mg/ml dexamethasone that will be injected in 5 ml aliquots after negative aspiration.The control group will receive 1 mL of normal saline.
  * After completion of the surgical procedure, a patient will be transferred to Post-Anesthesia Care Unit (PACU). Paracetamol 15 mg/kg IV will be administered every 6 hours after discharge to the ward.

ELIGIBILITY:
Inclusion Criteria:

* Patients, aged 21-75 years
* American Society of Anesthesiologists (ASA) physical status I-III
* Scheduled to undergo unilateral total hip replacement surgery.

Exclusion Criteria:

* Patient refusal.
* Known hypersensitivity to local anesthetics.
* Body mass index > 35 kg /m2.
* Uncooperative or psychiatric patients.
* Infection at the injection site.
* Coagulation disorder.
* Major cardiac, renal, or hepatic diseases

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Time for first request of rescue analgesia | The first day after surgery
  Time to the first call for morphine rescue analgesia.

SECONDARY OUTCOMES:
Postoperative morphine consumption | The first day after surgery
  Total morphine consumption (rescue analgesia) in the first day postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Abdelkhalik, M.D, Study Director — Assistant Professor of Anesthesia and Intensive Care, Tanta University
Locations (1):
- Tanta University, Tanta, Algharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Once the study had been successfully completed, the data will be shared with other researchers.
Supporting Information: Study Protocol, ICF
Time Frame: - Within 6 months from acceptance of publication
Access Criteria: samehabdelkhalik1982@gmail.com